CLINICAL TRIAL: NCT01230515
Title: Opioid Titration in the Hospice Setting: Barriers Assessment and Modification of the Model Order Sheet and Protocol
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC SUPP 0566; P30CA068485 (NIH)
Record Dates: First submitted 2010-10-11; First posted 2010-10-29 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Cancer Pain
Keywords: Oncology Pain Management in outpatient hospice setting
MeSH Terms: conditions — Cancer Pain | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Caregiver: Family members will be asked to complete a demographic survey, an assessment of the patient's current pain, and a series of questionnaires including: Caregiver Pain Medicine Questionnaire, the Stressful Caregiving Adult Reactions To Experiences of Dying Scale, and the Caregivers' Self Efficacy in Pain Management Questionnaire. Upon completion of the questionnaires, patients and caregivers will be interviewed separately.
  Interventions: Other: interview, focus group and structured survey
- Hospice staff: Hospice staff will be asked to complete the Pain Knowledge and Attitudes survey. They will also complete the Technology Acceptance Model (TAM) questionnaire to assess the perceived utility of an opioid titration order sheet to help manage pain control. A demographic survey will also be completed.
  Interventions: Other: interview, focus group and structured survey
- Referring physician: Referring physicians will be asked to complete the Pain Knowledge and Attitudes survey as well as the TAM questionnaire and Demographic Survey.
  Interventions: Other: interview, focus group and structured survey
- Patient: Demographic information includes education, marital status, number in household, and employment status will be obtained from patient. Clinical data will be obtained from the patient's medical records. Information to be obtained will include information about the type of cancer, stage of disease, time since diagnosis, current treatment for cancer, type of pain, time since onset of pain, and time of first opioid prescription. The patient will also take a pain assessment survey.
  Interventions: Other: Individual patient interview, focus group and structured survey

INTERVENTIONS:
Other: Individual patient interview, focus group and structured survey
  Groups: Patient
Other: interview, focus group and structured survey
  Groups: Caregiver
Other: interview, focus group and structured survey
  Groups: Hospice staff
Other: interview, focus group and structured survey
  Groups: Referring physician

SUMMARY:
The purpose of this study is to modify the opioid titration order sheet to meet the needs of the outpatient hospice population and to conduct a pilot trial to assess feasibility, utility, and derive preliminary efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility includes:

  * Alive Hospice outpatient
  * Diagnosis of carcinoma
  * Pain requiring fixed dose opioids
  * Age > 21 years
  * Not pregnant or lactating
  * Willing and able to sign informed consent
  * Able to speak/comprehend English

Caregiver eligibility will include:

* Caregiver for an Alive Hospice patient
* Willing and able to sign informed consent
* Able to speak/comprehend English

Hospice Staff eligibility will include:

* Currently on staff at Alive Hospice
* Willing and able to sign informed consent
* Able to read/speak English.

Referring Physician eligibility will include:

* Having recently referred patients to Alive Hospice
* Willing and able to sign informed consent and able to read/speak English.

Exclusion Criteria:

* patients < 21 years of age
* pregnant or lactating
* patients, caregiver and or Hospice staff that does not speak/comprehend English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospice Staff Caregiver Patient Referring Physician
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Adequate pain control | Until death.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingam Cancer Center, Nashville, Tennessee, United States